CLINICAL TRIAL: NCT03566511
Title: Use of Functional MRI to Assess Functional Hypothalamic Activation in Response to Diazoxide
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Grant funding ended. NIDDK grant renewed without an MR aim. No plans to do future studies.
Sponsor: Meredith Hawkins (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); American Diabetes Association (Other)
Responsible Party: Sponsor-Investigator, Meredith Hawkins, Principal Investigator, Albert Einstein College of Medicine
Organization: Albert Einstein College of Medicine (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2018-9040; R01DK069861 (NIH)
Record Dates: First submitted 2018-05-17; First posted 2018-06-25 (Actual); Results first posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus, Type 2; Glucose, High Blood; Glucose Metabolism Disorders (Including Diabetes Mellitus)
Keywords: diabetes; type 2 diabetes; insulin resistance; diazoxide; MRI
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Diabetes Mellitus; Insulin Resistance | interventions — Diazoxide

STUDY DESIGN:
Intervention Model Description: Study was initially intended to be a double blinded, randomized, crossover design; however, it was terminated early due to issues with magnetic resonance (MR) system.
Who Masked: Participant
Masking Description: The subject will be blinded to which study drug is received first (Drug or Placebo).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Healthy (Diazoxide) (Experimental): Proglycem, oral suspension (4-7 mg/kg). Healthy participants will receive diazoxide between MRI scans.
  Interventions: Drug: Diazoxide
- Healthy (Placebo) (Placebo Comparator): Taste-matched placebo. Healthy participants will receive placebo between MRI scans.
  Interventions: Drug: Placebo
- T2D (Diazoxide) (Experimental): Proglycem, oral suspension (4-7 mg/kg). Type 2 diabetic (T2D) participants will receive diazoxide between MRI scans.
  Interventions: Drug: Diazoxide
- T2D (Placebo) (Placebo Comparator): Taste-matched placebo. T2D participants will receive placebo between MRI scans.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diazoxide — Healthy and T2D participants will receive diazoxide at a dose of 4-7 mg/kg (based upon weight) between baseline MRI scan and second MRI scan.
  Other Names: Proglycem
  Arms: Healthy (Diazoxide); T2D (Diazoxide)
Drug: Placebo — Healthy and T2D participants will receive placebo between baseline MRI scan and second MRI scan.
  Arms: Healthy (Placebo); T2D (Placebo)

SUMMARY:
The goal of this study is to determine whether metabolic control centers in the brain can be activated in patients with type 2 diabetes (T2D) as compared to non-diabetic individuals. This is important since people with diabetes have inappropriately high production of glucose, which could be at least in part due to impaired activation of important brain centers.

DETAILED DESCRIPTION:
In this study investigators will use functional magnetic resonance imaging (fMRI), a safe, noninvasive method of measuring brain activity by imaging the blood flow to different parts of the brain, to assess the impact of the medication diazoxide on both diabetic and non-diabetic patients. fMRI is a technique for measuring and mapping brain activity. This technique relies on the fact that cerebral blood flow (CBF) and neuronal activity are coupled.

Previous rodent and human studies have demonstrated that diazoxide activates potassium (KATP) channels that are sensitive to ATP in the hypothalamus, inhibiting hepatic glucose production. However, these inhibitory effects of diazoxide on hepatic glucose production are curiously absent in diabetic patients, which suggests that they may have impaired activation of KATP channels and thus lowered brain activity in this area of the brain.

After screening and meeting eligibility criteria, participants will have 2 day-long study visits (one day in which the brain will be imaged before and after receiving diazoxide, and one day in which the brain will be imaged before and after placebo). Each study day will include up to 3 MRI scans per study visit and hourly blood draws.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes (T2D)

  * Age: Between 21 and 70 y.o.
  * BMI: <35
  * A1c 8.0-12.0%
  * Negative drug screen
  * Not suffering from proliferative retinopathy, significant diabetic renal disease or severe neuropathy (including cardiovascular and gastrointestinal autonomic dysfunction)
* Healthy (ND)

  * Age: Between 21 and 70 y.o.
  * BMI: <30
  * Negative drug screen
  * No family history of diabetes among first-degree relatives (mother, father)

Exclusion Criteria:

* Age: Under 21 or over 70 y.o.
* BMI: >35 for T2D and >30 for ND
* Hypertension
* Severe polydipsia and polyuria
* Uncontrolled hyperlipidemia
* Clinically significant liver dysfunction
* Clinically significant kidney dysfunction
* Anemia
* Clinically significant leukocytosis or leukopenia
* Clinically significant thrombocytopenia or thrombocytosis
* Coagulopathy
* Positive urine drug screen
* Urinalysis: Clinically significant abnormalities
* Clinically significant electrolyte abnormalities
* Smoking >10 cig/day
* Alcohol: Men >14 drinks/wk or > 4 drinks/day, Women >7 drinks/wk or >3 drinks/day
* History of chronic liver disease, active hepatitis infection, HIV/AIDS, chronic kidney disease (stage 3 or greater), active cancer, cardiovascular disease or other heart disease, systemic rheumatologic conditions, seizures, bleeding disorders, muscle disease
* Surgeries that involve removal of endocrine glands except for thyroidectomy
* Pregnant women
* Subject enrolled in another study less than one month prior to the anticipated start date of the proposed study
* Family history: family history of premature cardiac death
* Allergies to medication administered during study
* Uncontrolled psychiatric disorders
* Perimenopausal women who are experiencing/have experienced hot flashes
* Any contraindications for MRI: presence of any non-MRI compatible implants including pacemaker, aneurysm clip, cochlear implant, neurostimulator; history of eye injury with metal; history of ever being a metal worker; history of gunshot wounds or any other imbedded metal objects; history of claustrophobia or prior episodes of significant anxiety or discomfort while obtaining an MRI.
* Any condition which in the opinion of the PI makes the subject ill-suited for participation in the study

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Hawkins, M.D., M.S., Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 37 patients signed consent and were screened for eligibility. Following screening, 22 patients were deemed eligible. Of the 22, 11 did not enroll in the study after passing the screening for various reasons including being lost to follow-up or unable to commit. In summary, 11 patients were enrolled and randomized into the study; however, randomization order cannot be verified from documentation for 3 study patients. These 3 patients did not complete the overall study and were never unblinded.
Groups:
- Diazoxide First Then Matched Placebo: Proglycem, oral suspension (4-7 mg/kg). Healthy participants will receive Diazoxide between MRI scans.
  Diazoxide: Healthy participants will receive Diazoxide at a dose of 4-7 mg/kg (based upon body weight) between baseline MRI scan and second MRI scan.
  Matched placebo:
  Healthy participants will receive placebo between baseline MRI scan and second MRI scan.
- Matched Placebo First Then Diazoxide: Proglycem, oral suspension (4-7 mg/kg). T2D participants will receive Diazoxide between MRI scans.
  Diazoxide: T2D participants will receive Diazoxide at a dose of 4-7 mg/kg (based upon body weight) between baseline MRI scan and second MRI scan.
  Matched placebo:
  T2D participants will receive placebo between baseline MRI scan and second MRI scan.
Period: 1st Intervention (1 Day)
Arm/Group | Diazoxide First Then Matched Placebo | Matched Placebo First Then Diazoxide
Started | 4 | 4
Completed | 3 | 4
Not Completed | 1 | 0
Not completed — Study terminated and participant never received Diazoxide (DZX) | 1 | 0
Period: Washout (~1 Month)
Arm/Group | Diazoxide First Then Matched Placebo | Matched Placebo First Then Diazoxide
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0
Period: 2nd Intervention (1 Day)
Arm/Group | Diazoxide First Then Matched Placebo | Matched Placebo First Then Diazoxide
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: As described in the 'Participant Flow' module, 11 patients were enrolled and randomized into the study; however, randomization order could not be verified from documentation for 3 of the study patients. These 3 patients did not complete the overall study and were never unblinded.
Groups:
- All Study Participants: Proglycem, oral suspension (4-7 mg/kg). Healthy participants will receive Diazoxide between MRI scans.
  Diazoxide: Participants will receive Diazoxide at a dose of 4-7 mg/kg (based upon body weight) between baseline MRI scan and second MRI scan.
  Participants will receive placebo between baseline MRI scan and second MRI scan.
Arm/Group | All Study Participants
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Arterial Spin Labeling (ASL) Signal Measured Using 3T MRI From Baseline to 5 Hours Post Dosing
Description: Arterial Spin Labeling data was acquired and converted by the Gruss Magnetic Resonance Research Center (MRRC) and reported as Hypothalamic Cerebral Blood Flow (CBF) which is a more meaningful clinical endpoint measurement. Data was collected at three time points during each of the two study visits (pre dosing, 2 hours post dosing, and 5 hours post dosing). CBF values at the respective timepoints are summarized in mL/100g/min units and reported by study arm. An increase in CBF is correlated with an increase in brain activity.
Time Frame: 2 hours and 5 hours post dosing
Population: 7 patients were able to complete both studies within the crossover design as described in the 'Participant Flow' module and have their data analyzed. An additional 4 patients (3 healthy, and 1 T2D) were not able to complete their measurements and, therefore, no data are available for these patients. Standard error (SE) data for the DZX studies were derived from visual estimates of the bar graphs. SE data for the Placebo studies were extrapolated from DZX studies.
Measure: Mean (Standard Error); unit: mL/100g/min
Groups:
- Diazoxide: Proglycem, oral suspension (4-7 mg/kg). Healthy participants will receive Diazoxide between MRI scans.
  Diazoxide: Participants will receive Diazoxide at a dose of 4-7 mg/kg (based upon body weight) between baseline MRI scan and second MRI scan.
  Matched placebo:
  Participants will receive placebo between baseline MRI scan and second MRI scan.
- Matched Placebo: Proglycem, oral suspension (4-7 mg/kg). T2D participants will receive Diazoxide between MRI scans.
  Diazoxide: Participants will receive Diazoxide at a dose of 4-7 mg/kg (based upon body weight) between baseline MRI scan and second MRI scan.
  Matched placebo:
  Participants will receive placebo between baseline MRI scan and second MRI scan.
Arm/Group | Diazoxide | Matched Placebo
Number analyzed (Participants) | 7 | 7
mL/100g/min
  Baseline | 29.78 (1.3) | 28.36 (1.3)
  2 hours | 26.52 (1.7) | 26.25 (2.0)
  5 hours | 28.88 (1.4) | 27.75 (1.4)

ADVERSE EVENTS:
Time Frame: Two, 8-hour visits, up to one month apart
Arm/Group | Diazoxide | Matched Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diazoxide (N=7) | Matched Placebo (N=7)
Uncomfortable (General disorders) | 0 | 1 — Verbatim Term: Patient felt "hot and tired" inside the MRI machine.

LIMITATIONS AND CAVEATS:
Instrumentation got remodeled and further studies were unable to be conducted and the trial was unable to be completed as proposed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/11/NCT03566511/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/11/NCT03566511/ICF_001.pdf